CLINICAL TRIAL: NCT01546103
Title: Pilot Study of Vitamin D3 Supplementation and Outcomes in Vitamin D Deficient Obese, African American Adolescents
Brief Title: Vitamin D3 Supplementation Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-008075
Record Dates: First submitted 2012-01-04; First posted 2012-03-07 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 supplementation of 1000 IU (Active Comparator)
  Interventions: Dietary Supplement: Cholecalciferol
- Vitamin D3 supplementation of 5000 IU (Active Comparator)
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 1000 IU by mouth, once daily for 3 months.
  Other Names: Vitamin D
  Arms: Vitamin D3 supplementation of 1000 IU
Dietary Supplement: Cholecalciferol — 5000 IU by mouth, once daily for 3 months.
  Other Names: Vitamin D
  Arms: Vitamin D3 supplementation of 5000 IU

SUMMARY:
The purpose of this research study is to determine whether taking vitamin D, every day, over a 12 week period will improve the vitamin D status, risks for poor heart health, risks for developing type 2 diabetes, and/or muscle strength in overweight, African American teenagers with low vitamin D levels.

DETAILED DESCRIPTION:
Vitamin D deficiency/insufficiency is common throughout the lifespan, and across all race and ethnic groups. The American Academy of Pediatrics (AAP) recently recommended supplementation dose to 400 international units (IU) daily in all children. These recommendations target rickets prevention, but address neither the vitamin D supplementation necessary to optimize bone health nor the nontraditional vitamin D roles in immune disease, insulin resistance, muscle function, and cardiovascular disease (CVD). Moreover, the AAP recommendation noted that it had little pediatric data upon which to base guidelines. The Institute of Medicine also recently published Dietary Reference Intakes for Calcium and Vitamin D: the estimated average requirement in children and adults was set at 400(IU) daily and the recommend dietary allowance was set at 600 IU daily. Data on outcomes and supplementation levels in African Americans (a population at particular risk for vitamin D deficiency) and across pediatric age ranges and body habitus types, are lacking. The Vitamin D supplementation requirement in obese, African American adolescents is particularly problematic since obesity is associated with 1) lower circulating vitamin D levels (25OHD) and 2) insulin resistance. This pilot study will examine the effect of vitamin D supplementation upon 25OHD, the serum marker of vitamin D status, in obese, African American adolescents with vitamin D deficiency. Subjects will be randomized to receive cholecalciferol 1000 IU or 5000 IU daily for 3 months. Serum 25OHD, parathyroid hormone, glucose, insulin, CVD risk markers, and measures of muscle function and pain will be obtained at baseline and post-treatment. This pilot study will provide data on serum 25OHD responses to vitamin D at doses more likely to meaningfully impact 25OHD than the current American Academy of Pediatrics (AAP) supplementation guideline. Responses to supplementation can then inform future clinical trials aimed at addressing outcomes of vitamin D replacement on insulin sensitivity and CVD risk in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Obese [body mass index (BMI) greater than or equal to 95th percentile for age and sex]
* Pubertal (Tanner Stage greater than 1)
* 25OHD less than 20 ng/mL (for treatment phase); if 25OHD is greater than or equal to 20 ng/mL, only baseline data will be obtained.
* Committed to adherence to supplementation and study completion

Exclusion Criteria:

* Pregnancy
* Chronic medical conditions or medications use that can affect growth, nutrition, bone health, vitamin D metabolism, glucose, or insulin sensitivity
* Known history of hypercalcemia or hypercalciuria
* Non-English speaking, as assessments are available only in English

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Serum 25OHD before and after treatment | 12 weeks
  The analysis will be an intention-to-treat method in which subjects are assumed to obtain all vitamin D supplements from the study and from no other sources, and all subjects are assumed to comply with their assigned dose and daily use. For the main contrasts of interest (5000 IU vs 1000 IU doses as well as serum 25OHD concentrations), we propose a longitudinal mixed effects model with time measurements at 0 and 12 weeks.

SECONDARY OUTCOMES:
Adiponectin level comparison | 12 weeks
  Adiponectin level comparison before and at post-treatment
Lipid panel comparison | 12 weeks
  Lipid panel comparison before and at post-treatment
Lipoprotein subclass particles comparison | 12 weeks
  Lipoprotein subclass particles comparison before and at post-treatment
High-sensitivity C-Reactive Protein (hsCRP) comparison | 12 weeks
  High-sensitivity C-Reactive Protein (hsCRP) comparison before and at post-treatment
Insulin level comparison | 12 weeks
  Insulin level comparison before and at post-treatment
Total and undercarboxylated osteocalcin level comparison | 12 weeks
  Total and undercarboxylated osteocalcin level comparison before and at post-treatment
Muscle strength comparison | 12 weeks
  Muscle strength comparison before and at post-treatment
Musculoskeletal pain comparison | 12 weeks
  Musculoskeletal pain comparison before and at post-treatment
Blood pressure comparison | 12 weeks
  Blood pressure comparison before and at post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sheela N Magge, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Andrea Kelly, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States